CLINICAL TRIAL: NCT02185820
Title: A MULTICENTER, OPEN LABEL PHASE I/II STUDY OF CARFILZOMIB, POMALIDOMIDE AND DEXAMETHASONE IN RELAPSED AND/OR REFRACTORY MULTIPLE MYELOMA (MM) PATIENTS
Brief Title: Phase I/II Study of Carfilzomib, Pomalidomide and Dexamethasone in Relapsed And/Or Refractory Multiple Myeloma Patients (CPD)
Acronym: CPD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: European Myeloma Network B.V. (Network)
Collaborators: University of Turin, Italy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMN07/IST-CAR-538
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Relapsed and/or refractory; CPD
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Treatment schedule for 8 cycles of induction:
  Carfilzomib = 20 mg/m2 IV once daily on days 1 of cycle 1 only followed by 27/36/45/56 mg/m2 days 8, 15 in cycle 1, then for all subsequent doses 27/36/45/56 mg/m2 IV once daily on days 1, 8, 15 followed by 13-day rest period (day 16 through 28).
  Pomalidomide = 4 mg daily on days 1 - 21 every 28 days. Dexamethasone = 20 mg on days 1, 8, 15, 22 every 28 days.
  Treatment schedule for maintenance until progression or intolerance:
  Carfilzomib = at the MTD achieved in the phase I of the study on days 1, 8, 15 in 28-days cycles.
  Pomalidomide = 4 mg daily on days 1 - 21 every 28 days. Dexamethasone = 20 mg on days 1, 8, 15, 22.
  Interventions: Drug: Carfilzomib; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib
Drug: Pomalidomide
Drug: Dexamethasone

SUMMARY:
This protocol is a phase I/II multicenter study designed to assess the safety and the efficacy of the proposed combinations in relapsed and/or refractory Multiple Myeloma (MM) patients.

DETAILED DESCRIPTION:
TREATMENT PERIOD Patients will start the salvage treatment with CPd, as soon as the screening visits of the pre-treatment period have been terminated. Patients will receive 8 CPd cycles.

PHASE I

In the phase I part of the study, the following dose levels of pomalidomide will be studied with a constant dose of dexamethasone and carfilzomib:

Level -1 Carfilzomib = 20 mg/m2 IV once daily on days 1 of cycle 1 only followed by 27 mg/m2 days 8, 15 in cycle 1, then for all subsequent doses 27 mg/m2 IV once daily on days 1, 8, 15 followed by 13-day rest period (day 16 through 28).

Pomalidomide = 4 mg daily on days 1 - 21 every 28 days. Dexamethasone = 20 mg on days 1, 8, 15, 22 every 28 days. Level 0 (starting dose) Carfilzomib = 20 mg/m2 IV once daily on days 1 of cycle 1 only followed by 36 mg/m2 days 8, 15 in cycle 1, then for all subsequent doses 36 mg/m2 IV once daily on days 1, 8, 15 followed by 13-day rest period (day 16 through 28).

Pomalidomide = 4 mg daily on days 1 - 21 every 28 days. Dexamethasone = 20 mg on days 1, 8, 15, 22 every 28 days. Level +1 Carfilzomib = 20 mg/m2 IV once daily on days 1 of cycle 1 only followed by 45 mg/ m2 days 8, 15 in cycle 1, then for all subsequent doses 45 mg/m2 IV once daily on days 1, 8, 15 followed by 13-day rest period (day 16 through 28).

Pomalidomide = 4 mg daily on days 1 - 21 every 28 days. Dexamethasone = 20 mg on days 1, 8, 15, 22 every 28 days. Level +2 Carfilzomib = 20 mg/m2 IV once daily on days 1 of cycle 1 only followed by 56 mg/m2 days 8, 15 in cycle 1, then for all subsequent doses 56 mg/m2 IV once daily on days 1, 8, 15 followed by 13-day rest period (day 16 through 28).

Pomalidomide = 4 mg daily on days 1 - 21 every 28 days. Dexamethasone = 20 mg on days 1, 8, 15, 22 every 28 days. Patients will be observed during the first cycle of therapy for the assessment of side effects and observation of DLTs.

Dose escalation will proceed as follows:

3 patients will be entered at dose level 0. If none of the 3 experience DLT, dose escalation will continue. If one of three patients experience DLT, three additional patients will be added to this cohort (max 6).

If two of three patients experience a DLT at any given dose, the MTD will have been exceeded and the MTD will be the preceding dose at which < one of 6 patients experienced a DLT.

If no further patients experience DLT (1 of 6) dose escalation will continue. If 2 patients experience DLT (2 of 6) the MTD will have been exceeded and the MTD will be the previous dose at which <1 patient of 6 experienced DLT.

The phase I of the study will end once the MTD has been defined.

PHASE II The phase II of the study will start after the MTD has been defined in the phase I of the study. The dose used to treat patients in the phase II will be the MTD defined in the phase I of the study.

In the second part of the study, the MTD of the association CPd (or in absence of any MTD observed) the doses of dose level 3 (maximum per protocol dose) will be administered to a total of 45 consecutive patients in order to assess response rate and clinical efficacy.

THE PHASE 2 OF THE STUDY WILL START ONLY AFTER THE ANALYSIS OF THE PHASE 1 RESULTS AND THE RELEVANT STUDY REPORT.

MANTEINANCE PERIOD

At the end of 8 courses, maintenance phase will start. Patients will receive:

Carfilzomib = at the MTD achieved in the phase I of the study on days 1, 8, 15 in 28-days cycles.

Pomalidomide = 4 mg daily on days 1 - 21 every 28 days. Dexamethasone = 20 mg on days 1, 8, 15, 22. Patients will be stopped at PD or intolerance. For the maintenance period a continuous assessment of the toxicity and tolerability profile of the CPd combination could permit to the Investigators to continue the treatment using Pomalidomide or Carfilzomib alone according to the dose modification plan.

ELIGIBILITY:
Inclusion Criteria:

Age > 18 years. Eastern Cooperative Oncology Group (ECOG) performance status 0-2. Patient is, in the investigator(s) opinion, willing and able to comply with the protocol requirements.

Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.

Female patient is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.

Male patient agrees to use an acceptable method for contraception (i.e., condom or abstinence) for the duration of the study.

Patients who are primary refractory or relapsed/refractory to Lenalidomide. Subjects must have been received at least 2 consecutive cycles of a prior treatment that include Lenalidomide alone or in combination.

Subject must be primary refractory or relapsed/refractory to Lenalidomide, defined as: 1) never achieved any response better than progressive disease (PD) to any Lenalidomide-containing regimen; 2) documented disease progression during or within 60 days of completing their last myeloma Lenalidomide-containing regimen.

Both relapsed and/or refractory to Bortezomib and naive to Bortezomib patients can be enrolled.

Patient has measurable disease, defined as follows: any quantifiable serum monoclonal protein value (generally, but not necessarily, ≥ 0.5 g/dL of M-protein) and, where applicable, urine light-chain excretion of >200 mg/24 hours. For patients with oligo or non-secretory MM, it is required that they have measurable plasmacytoma > 2 cm as determined by clinical examination or applicable radiographs (i.e. MRI, CT-Scan) or an abnormal free light chain ratio (n.v.: 0.26-1.65). We anticipate that less than 10% of patients admitted to this study will be oligo- or non-secretory MM with free light chains only in order to maximize interpretation of benefit results.

Patient has a Karnofsky performance status ≥60%. Patient has a life-expectancy >3 months.

Patient has the following laboratory values within 14 days before Baseline (day 1 of the Cycle 1, before study drug administration):

Platelet count ≥ 50 x 109/L (≥ 30 x 109/L if myeloma involvement in the bone marrow is > 50%) within 14 days prior to drug administration).

Hemoglobin ≥ 8 g/dL (80 g/L) within 14 days prior to enrollment (subjects may be receiving red blood cell [RBC] transfusions in accordance with institutional guidelines).

Absolute neutrophil count (ANC) ≥ 1 x 109/L without the use of growth factors. Corrected serum calcium ≤14 mg/dL (3.5 mmol/L) Alanine transaminase (ALT): ≤ 3.5 x the ULN. Total bilirubin: ≤ 2 x the ULN. Calculated or measured creatinine clearance ≥ 45 mL/min.

Exclusion Criteria:

Newly diagnosed myeloma patients. Patient with non-secretory MM, unless serum free light chains are present and the ratio is abnormal.

Pregnant or lactating females. Major surgery within 21 days prior to enrollment. Acute active infection requiring treatment (systemic antibiotics, antivirals, or antifungals) within 14 days prior to enrolment.

Patient has active infectious hepatitis type A, B or C or HIV. Unstable angina or myocardial infarction within 4 months prior to enrollment, NYHA Class III or IV heart failure, uncontrolled angina, history of severe coronary artery disease, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or Grade 3 conduction system abnormalities unless subject has a pacemaker.

Uncontrolled hypertension or uncontrolled diabetes within 14 days prior to enrollment.

Significant neuropathy (Grades 3-4, or Grade 2 with pain) within 14 days prior to enrollment.

Known history of allergy to Captisol (a cyclodextrin derivative used to solubilize carfilzomib).

Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to all anticoagulation and antiplatelet options, antiviral drugs, or intolerance to hydration due to pre-existing pulmonary or cardiac impairment.

Subject with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to baseline.

Any other clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent.

Nonhematologic malignancy within the past 3 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason Grade 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal or pancreas.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
DLT | 1 year
  The dose-limiting toxicity (DLT) and maximum tolerated dose (MTD) of carfilzomib, pomalidomide and dexamethasone (CPd) association.
Partial response | 3 years
  Determine the rate of partial response (PR) with the CPd association: a PR rate of 25% (p0) is considered not promising (H0) and a 45% (p1) as interesting.

SECONDARY OUTCOMES:
Toxicities | 3 years
  Less than 30% of patients presenting the following toxicities: grade 4 neutropenia lasting > 1 week, any grade 4 hematological toxicities except neutropenia, any > grade 3 extra-hematologic toxicities.
PFS | 3 years
  Determine the progression-free survival (PFS).
TTP | 3 years
  Determine the time to progression (TTP).
DFS | 3 years
  Determine the disease free survival (DFS).
DOR | 3 years
  Determine the duration of response (DOR).
TTNT | 3 years
  Determine the time to next therapy (TTNT).
OS | 3 years
  Determine the overall survival (OS).
Tumor response and survival | 3 years
  Determine whether tumor response and survival might significantly change in particular subgroups of patients defined on prognostic factors (β2-microglobulin, C-reactive protein (CRP), FISH).

CONTACTS AND LOCATIONS:
Overall Officials: Sara Bringhen, MD, Principal Investigator — A.O.U. Città della Salute e della Scienza
Locations (1):
- Dipartimento di Biotecnologie Molecolari e Scienze per la Salute, Torino, Italy